CLINICAL TRIAL: NCT06708286
Title: A Randomized, Blinded, Controlled Clinical Trial to Evaluate the Immunogenicity and Safety of Adsorbed Cell-free DTP Vaccine (Five-component)
Brief Title: A Clinical Trials of Adsorbed Cell-free DPT Vaccine (Five-component)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-Tdcp-002
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-11

CONDITIONS: Diphtheria; Tetanus; Pertussis
Keywords: Vaccine; Five Components; Immunogenicity; Safety; Acellular
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough | interventions — Tetanus Toxoid; Vaccines, Combined; Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Phase II, ≥18 years old, Experimental vaccine (Experimental): One dose of Tdcp on Day 0
  Interventions: Biological: Tetanus, Reduced Diphtheria and Acellular Pertussis (Five Components) Combined Vaccine, Adsorbed (Tdcp))
- Phase II, ≥18 years old, Control vaccine (Active Comparator): One dose of PPV23 on Day 0
  Interventions: Biological: 23-valent Pneumococcal Polysaccharide Vaccine (PPV23)
- Phase II, 7-17 years old, Experimental vaccine (Experimental): One dose of Tdcp on Day 0
  Interventions: Biological: Tdcp
- Phase II, 7-17 years old, Control vaccine (Active Comparator): One dose of PPV23 on Day 0
  Interventions: Biological: PPV23
- Phase III, ≥18 years old, Experimental vaccine (Experimental): One dose of Tdcp on Day 0
  Interventions: Biological: Tdcp
- Phase III, ≥18 years old, Control vaccine (Active Comparator): One dose of PPV23 on Day 0
  Interventions: Biological: PPV23
- Phase III, 7-17 years old, Experimental vaccine (Experimental): One dose of Tdcp on Day 0
  Interventions: Biological: Tdcp
- Phase III, 7-17 years old, Control vaccine (Active Comparator): One dose of PPV23 on Day 0
  Interventions: Biological: PPV23
- Phase III, 6 years old, Experimental vaccine (Experimental): One dose of Tdcp on Day 0
  Interventions: Biological: Tdcp
- Phase III, 6 years old, Control vaccine (Active Comparator): One dose of DTaP on Day 0
  Interventions: Biological: Diphtheria-tetanus-acellular pertussis vaccine (DTaP)

INTERVENTIONS:
Biological: Tetanus, Reduced Diphtheria and Acellular Pertussis (Five Components) Combined Vaccine, Adsorbed (Tdcp)) — 1 dose of Tdcp vaccine (0.5ml) on day 0
  Arms: Phase II, ≥18 years old, Experimental vaccine
Biological: 23-valent Pneumococcal Polysaccharide Vaccine (PPV23) — 1 dose of PPV23 vaccine (0.5ml) on day 0
  Arms: Phase II, ≥18 years old, Control vaccine
Biological: Tdcp — 1 dose of Tdcp vaccine (0.5ml) on day 0
  Arms: Phase II, 7-17 years old, Experimental vaccine
Biological: PPV23 — 1 dose of PPV23 vaccine (0.5ml) on day 0
  Arms: Phase II, 7-17 years old, Control vaccine
Biological: Tdcp — 1 dose of Tdcp vaccine (0.5ml) on day 0
  Arms: Phase III, ≥18 years old, Experimental vaccine
Biological: PPV23 — 1 dose of PPV23 vaccine (0.5ml) on day 0
  Arms: Phase III, ≥18 years old, Control vaccine
Biological: Tdcp — 1 dose of Tdcp vaccine (0.5ml) on day 0
  Arms: Phase III, 7-17 years old, Experimental vaccine
Biological: PPV23 — 1 dose of PPV23 vaccine (0.5ml) on day 0
  Arms: Phase III, 7-17 years old, Control vaccine
Biological: Tdcp — 1 dose of Tdcp vaccine (0.5ml) on day 0
  Arms: Phase III, 6 years old, Experimental vaccine
Biological: Diphtheria-tetanus-acellular pertussis vaccine (DTaP) — 1 dose of DTaP vaccine (0.5ml) on day 0
  Arms: Phase III, 6 years old, Control vaccine

SUMMARY:
This is a randomized, blinded, controlled phase II and III clinical trial evaluating the immunogenicity and safety of adsorbed cell-free DPT vaccine. 320 subjects aged 7 years and older in the phase II were divided into two age groups, the ≥18 years group and the 7-17 years group, and randomized 3:1 to receive the trial vaccine Tdcp versus the control vaccine PPV23. 1500 subjects in the phase III were divided into 3 age subgroups. 780 subjects were planned to be enrolled in the 6-year-old group and randomized 1:1 to receive the experimental vaccine Tdcp versus the control vaccine DTaP, and 360 subjects were planned to be enrolled in each of the 7-17 and ≥18 age groups and randomized 3:1 to receive the experimental vaccine Tdcp versus the control vaccine PPV23.

ELIGIBILITY:
Inclusion Criteria:

* Phase II : People ≥ 7 years old
* Phase II : Willing to provide identification documents
* Phase II : Volunteers must obtain informed consent from the volunteers themselves and/or their guardians/ or delegates, sign the informed consent form and be willing to comply with the requirements of the clinical trial protocol, and be able to complete the full study follow-up
* Phase II : Volunteers aged 7~11 years have completed 4 doses of vaccine containing DPT
* Phase II : ≥12 years old volunteers need to have not received any component vaccine containing DPT within 5 years
* Phase III : People ≥6 years old
* Phase III : Willing to provide identification documents
* Phase III : Volunteers must obtain informed consent from themselves and/or their guardians/ or delegates, sign the informed consent form and be willing to comply with the requirements of the clinical trial protocol, and be able to complete the full study follow-up
* Phase III : Volunteers aged 6~11 years old have completed 4 doses of DPT-containing vaccine in the past
* Phase III : Volunteers aged ≥12 years should not have received any vaccine containing any component of DPT within 5 years

Exclusion Criteria:

* Those who have fever before vaccination, with axillary temperature >37.0℃;
* Females with a positive urine pregnancy test or breastfeeding volunteers, volunteers or their partners who have a pregnancy plan within 6 months;
* Suffering from hypertension (systolic blood pressure ≥160mmHg, diastolic blood pressure ≥100mmHg) that cannot be controlled by medication (applicable to people aged 18 years and above);
* Those who have already suffered from one of the diphtheria or tetanus diseases, those who have suffered from whooping cough in the last 3 years; or those who have had persistent cough for 14 days or more in the last 6 months;
* Those who have received vaccine containing pneumococcal polysaccharide/conjugate component within 5 years (applicable to those aged 7 years and above);
* Individuals who have had household contact with an individual with a confirmed diagnosis of pertussis, diphtheria, or tetanus disease in the past 30 days;
* Individuals who are allergic to the components of the test vaccine (e.g., aluminum adjuvant, sodium dihydrogen phosphate, sodium chloride, etc.) or who have developed an allergy to the same type of vaccine previously; individuals with a previous history of severe allergy, e.g., recurrent generalized urticaria, anaphylactic shock, respiratory distress, angioneurotic edema, or a history of asthma;
* Those with encephalopathy, uncontrolled epilepsy and other progressive neurological disorders (e.g., transverse myelitis, Guillain-Barre syndrome, demyelinating diseases)
* Persons with primary and secondary impaired immune function, receiving immunosuppressive therapy
* Doctor-diagnosed coagulation abnormalities (e.g. coagulation factor deficiencies, coagulopathies, platelet abnormalities) or significant bruising or coagulation disorders
* Currently suffering from severe chronic diseases, acute exacerbation of chronic diseases, acute infectious diseases;
* Have received another investigational drug or vaccine within 1 month prior to receiving the experimental vaccine, or have plans to participate or are participating in a clinical study of any other drug;
* Have received an injectable live attenuated vaccine within 14 days prior to receiving the experimental vaccine, or any other vaccine within 7 days prior to receiving the experimental vaccine;
* In the judgment of the investigator, the volunteer has any other factors that make him/her unsuitable for participation in the clinical trial.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1820 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Phase II: Incidence of adverse reactions | Within 0-30 days after vaccination
Phase III: Geometric mean concentration (GMC) of serum anti-PT, FHA, PRN, FIM 2&3, DT, TT antibodies | Pre-vaccination and 30 days post-vaccination
Phase III: Proportion of serum anti-DT and TT antibodies ≥ 0.1IU/ml | 30 days after vaccination
Phase III: Incidence of adverse reactions | Within 0-30 days after vaccination

SECONDARY OUTCOMES:
Phase II: Incidence of adverse events/reactions | Within 30 minutes of vaccination
Phase II: Incidence of adverse events/reactions | 0-7 days after vaccination
Phase II: Incidence of adverse events | 0-30 days after vaccination
Phase II: Incidence of serious stadverse events | Within 6 months of vaccination
Phase III: Positive rate of serum anti-Pertussis Toxoid (PT), Filamentous hemagglutmin (FHA), Pertactin (PRN), FIM 2&3, Diphtheria Toxoid (DT), Tetanus Toxoid (TT) antibodies | 30 days after vaccination
Phase III: Positive transfer rate of serum anti-PT, FHA, PRN, FIM 2&3, DT, TT antibodies | 30 days after vaccination
Phase III: Geometric Mean Increase (GMI) of serum anti-PT, FHA, PRN, FIM 2&3, DT, TT antibodies | 30 days after vaccination
Phase III: Incidence of adverse events/reactions | Within 30 minutes of vaccination
Phase III: Incidence of adverse events/reactions | 0-7 days after vaccination
Phase III: Incidence of adverse events | 0-30 days after vaccination
Phase III: Incidence of SAEs in subjects aged 7 years and older | Within 6 months of vaccination
Phase III: Incidence of SAEs in subjects aged 6 years | Within 12 months of vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Hanqing He, Principal Investigator — Ethical Review Committee for Clinical Trials of Zhejiang Center for Disease Control and Prevention
Locations (1):
- Kaihua County Center for Disease Control and Prevention, Kaihua, China